CLINICAL TRIAL: NCT04002570
Title: Effects of Adjuvant Radiotherapy on Bone-marrow Derived and Immune Cells in Breast Cancer Patients
Brief Title: Adjuvant Radiotherapy on Circulating Cells in Breast Cancer Patients
Acronym: CCB-RT
Status: Completed | Type: Observational
Sponsor: Clinica Luganese Moncucco (Other)
Collaborators: Curzio Rüegg, MD, Head of Department, University of Fribourg (Unknown); Swiss National Science Foundation (Other); Tsoutsou Pelagia MD, Head of Radation Therapy Department (Unknown)
Responsible Party: Principal Investigator, Alessandra Franzetti Pellanda, Head of Radiation Therapy, Clinica Luganese Moncucco
Other Study IDs: CirculatingCellsBreast-RT
Record Dates: First submitted 2019-06-25; First posted 2019-06-28 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: breast cancer; circulating bone marrow-derived cells; circulating immune cells; radiotherapy; conservative treatment; disease control
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- GROUP I/GROUP I bis: 20 breast cancer patients who performed radiotherapy treatment
  Interventions: Other: blood samples collection
- GROUP II: maximum 10 patients who performed radiotherapy and chemotherapy and/or immunotherapy and/or neo-adjuvant hormone therapy or/and adjuvant immunotherapy/hormone therapy.
  Interventions: Other: blood samples collection
- CONTROLS GROUP: healthy women with +/- 5 years compared to breast cancer patients age
  Interventions: Other: blood samples collection

INTERVENTIONS:
Other: blood samples collection — blood samples collection are performed at 4 different timepoints: preop, pre rt, week 6 rt, week 12-14 (fu) for GROUP I and GROUP II; blood samples collection are performed at 3 different timepoints: pre rt, week 6 rt, week 12-14 (fu) for GROUP I bis; blood samples collection are performed just once for control GROUP.

SUMMARY:
Radiation applied to the preserved breast during radiotherapy treatment activates numerous molecular cascades in tumor bed adjacent cells causing an inflammatory state. During this process, pre-clinical studies demonstrated CD11b + and CD11b+cKit+cells mobilization in the blood. These cells are involved in numerous processes during tumor progression/control and metastases development. The expected results in clinical setting allow us to investigate the development of innovative therapeutic and monitoring strategies. The clinical repercussions would consist in identifying new predictive and prognostic targets in breast cancer.

DETAILED DESCRIPTION:
Every year, around one million women are newly diagnosed with breast cancer. Early screening and adjuvant treatments with curative intent such as radiotherapy, hormone therapy, chemotherapy, immunotherapy, have reduced the incidence of breast cancer specific mortality. Despite this, breast cancer remains the main cause of cancer mortality in Europe. The primary cause is due to metastases development in different organs, such as lung, liver, bones and brain. A significant decrease in mortality in breast cancer patients is likely to be achieved by preventing the formation of metastases or by implementing the efficacy of their treatment. Radiotherapy is one of the pillars of breast cancer adjuvant treatments with important survival benefits.

Mutual and dynamic communications between tumor cells and the tumor microenvironment (TME) influence the development and evolution of the tumor as well as the appearance of distant metastases. The mediators of the immune and inflammatory response that constitute TME, as well as mediators of tumor progression, are also considered "targets" of future therapeutic strategies.

Radiation applied to the preserved breast during radiotherapy treatment activates numerous molecular cascades in tumor bed adjacent cells causing an inflammatory state. During this process, pre-clinical studies demonstrated CD11b + and CD11b+cKit+cells mobilization in the blood. These cells are involved in numerous processes during tumor progression/control and metastases development. The results allow us to investigate the development of innovative therapeutic and monitoring strategies. The clinical repercussions would consist in identifying new predictive and prognostic targets in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer diagnosis bioptically proven with pre-operative clinical stage cT1-4, N0-1, M0;
* patients who are candidates for conservative surgery (tumorectomy / quadrantectomy +/- lymphadenectomy or sentinel lymph node) or patients already undergoing conservative surgery;
* patients who are candidates for an adjuvant mammary radiotherapy treatment +/- adjuvant or neoadjuvant chemotherapy due to a triple negative or a high ki67 value that has indicated it;
* understanding of the Italian language for the Coordinating Center, understanding of the French language for the satellite center.

Exclusion Criteria:

* previous mastectomy surgery;
* concomitant cancer diseases;
* previous chemo / radiotherapy treatments in the last three years.

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: patients performing treatments for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-10-25 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
the frequency of CD11b⁺cKit⁺ cells in peripheral blood and/or gene expression in circulating CD11b⁺ cells | pre surgery
  validate the hypothesis that adjuvant radiotherapy in breast cancer modulates the frequency of CD11b⁺cKit⁺ cells in peripheral blood and / or gene expression in circulating CD11b⁺ cells, evaluating their trend at different time points compared to radiotherapy treatment.
the frequency of CD11b⁺cKit⁺ cells in peripheral blood and/or gene expression in circulating CD11b⁺ cells | pre radiotherapy
  validate the hypothesis that adjuvant radiotherapy in breast cancer modulates the frequency of CD11b⁺cKit⁺ cells in peripheral blood and / or gene expression in circulating CD11b⁺ cells, evaluating their trend at different time points compared to radiotherapy treatment.
the frequency of CD11b⁺cKit⁺ cells in peripheral blood and/or gene expression in circulating CD11b⁺ cells | week 6 of radiotherapy
  validate the hypothesis that adjuvant radiotherapy in breast cancer modulates the frequency of CD11b⁺cKit⁺ cells in peripheral blood and / or gene expression in circulating CD11b⁺ cells, evaluating their trend at different time points compared to radiotherapy treatment.

SECONDARY OUTCOMES:
radiotherapy alters in a potentially predictive way the frequency of CD11b⁺cKit⁺ cells in peripheral blood | week 12-14 (fu)
  validate the hypothesis that adjuvant radiotherapy alters in a potentially predictive way the frequency of CD11b⁺cKit⁺ cells in peripheral blood and / or gene expression in circulating CD11b⁺ cells.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Franzetti Pellanda, MD, Principal Investigator — Clinica Luganese Moncucco
Locations (1):
- Clinica Luganese Moncucco, Lugano, Canton Ticino, Switzerland

REFERENCES:
- [Background] Ruegg CR, Chiquet-Ehrismann R, Alkan SS. Tenascin, an extracellular matrix protein, exerts immunomodulatory activities. Proc Natl Acad Sci U S A. 1989 Oct;86(19):7437-41. doi: 10.1073/pnas.86.19.7437. PMID 2477841
- [Background] Lorusso G, Ruegg C. The tumor microenvironment and its contribution to tumor evolution toward metastasis. Histochem Cell Biol. 2008 Dec;130(6):1091-103. doi: 10.1007/s00418-008-0530-8. Epub 2008 Nov 6. PMID 18987874
- [Background] Hanahan D, Coussens LM. Accessories to the crime: functions of cells recruited to the tumor microenvironment. Cancer Cell. 2012 Mar 20;21(3):309-22. doi: 10.1016/j.ccr.2012.02.022. PMID 22439926
- [Background] Coussens LM, Werb Z. Inflammation and cancer. Nature. 2002 Dec 19-26;420(6917):860-7. doi: 10.1038/nature01322. PMID 12490959
- [Background] Schlaeppi M, Ruegg C, Tran-Thang C, Chapuis G, Tevaearai H, Lahm H, Sordat B. Role of integrins and evidence for two distinct mechanisms mediating human colorectal carcinoma cell interaction with peritoneal mesothelial cells and extracellular matrix. Cell Adhes Commun. 1997 Mar;4(6):439-55. doi: 10.3109/15419069709004460. PMID 9177905
- [Background] Boylan AM, Ruegg C, Kim KJ, Hebert CA, Hoeffel JM, Pytela R, Sheppard D, Goldstein IM, Broaddus VC. Evidence of a role for mesothelial cell-derived interleukin 8 in the pathogenesis of asbestos-induced pleurisy in rabbits. J Clin Invest. 1992 Apr;89(4):1257-67. doi: 10.1172/JCI115710. PMID 1556187
- [Background] Ruegg C, Pytela R, Erle DJ. Characterization of the leukocyte integrin subunit beta 7. Chest. 1993 Feb;103(2 Suppl):86S. doi: 10.1378/chest.103.2_supplement.86s. No abstract available. PMID 8428547
- [Background] Sharma P, Sahni NS, Tibshirani R, Skaane P, Urdal P, Berghagen H, Jensen M, Kristiansen L, Moen C, Sharma P, Zaka A, Arnes J, Sauer T, Akslen LA, Schlichting E, Borresen-Dale AL, Lonneborg A. Early detection of breast cancer based on gene-expression patterns in peripheral blood cells. Breast Cancer Res. 2005;7(5):R634-44. doi: 10.1186/bcr1203. Epub 2005 Jun 14. PMID 16168108
- [Background] Kuonen F, Secondini C, Ruegg C. Molecular pathways: emerging pathways mediating growth, invasion, and metastasis of tumors progressing in an irradiated microenvironment. Clin Cancer Res. 2012 Oct 1;18(19):5196-202. doi: 10.1158/1078-0432.CCR-11-1758. Epub 2012 Jun 22. PMID 22730447
- [Background] Drooger JC, Hooning MJ, Seynaeve CM, Baaijens MH, Obdeijn IM, Sleijfer S, Jager A. Diagnostic and therapeutic ionizing radiation and the risk of a first and second primary breast cancer, with special attention for BRCA1 and BRCA2 mutation carriers: a critical review of the literature. Cancer Treat Rev. 2015 Feb;41(2):187-96. doi: 10.1016/j.ctrv.2014.12.002. Epub 2014 Dec 8. PMID 25533736
- [Background] Ruegg C, Yilmaz A, Bieler G, Bamat J, Chaubert P, Lejeune FJ. Evidence for the involvement of endothelial cell integrin alphaVbeta3 in the disruption of the tumor vasculature induced by TNF and IFN-gamma. Nat Med. 1998 Apr;4(4):408-14. doi: 10.1038/nm0498-408. PMID 9546785
- [Background] Han M, Liew CT, Zhang HW, Chao S, Zheng R, Yip KT, Song ZY, Li HM, Geng XP, Zhu LX, Lin JJ, Marshall KW, Liew CC. Novel blood-based, five-gene biomarker set for the detection of colorectal cancer. Clin Cancer Res. 2008 Jan 15;14(2):455-60. doi: 10.1158/1078-0432.CCR-07-1801. Epub 2008 Jan 18. PMID 18203981
- [Background] Coates AS, Winer EP, Goldhirsch A, Gelber RD, Gnant M, Piccart-Gebhart M, Thurlimann B, Senn HJ; Panel Members. Tailoring therapies--improving the management of early breast cancer: St Gallen International Expert Consensus on the Primary Therapy of Early Breast Cancer 2015. Ann Oncol. 2015 Aug;26(8):1533-46. doi: 10.1093/annonc/mdv221. Epub 2015 May 4. PMID 25939896
- [Background] Directive 2001/20/EC of the European Parliament and of the Council of 4 April 2001 on the approximation of the laws, regulations and administrative provisions of the member states relating to the implementation of good clinical practice in the conduct of clinical trials on medicinal products for human use. Med Etika Bioet. 2002 Spring-Summer;9(1-2):12-9. No abstract available. PMID 16276663
- [Background] Dixon JR Jr. The International Conference on Harmonization Good Clinical Practice guideline. Qual Assur. 1998 Apr-Jun;6(2):65-74. doi: 10.1080/105294199277860. PMID 10386329
- [Background] [The Helsinki Declaration of the World Medical Association (WMA). Ethical principles of medical research involving human subjects]. Pol Merkur Lekarski. 2014 May;36(215):298-301. No abstract available. Polish. PMID 24964504